CLINICAL TRIAL: NCT06746025
Title: Study of Newly Developed Program Designed to Create Greater Long-term Smoking Cessation Results.
Brief Title: Examining the Efficacy of a Newly Developed Smoking Cessation Program
Acronym: ESCaPe
Status: Completed | Type: Observational
Sponsor: Quit Center LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 052024CESS
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Nicotine Addiction; Smoking Cessation
Keywords: smoking; quit smoking; addiction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Session 1: Approximately 15-20 participants that have selected Session 1 as their preferred session
  Interventions: Behavioral: Quit Center cessation program

INTERVENTIONS:
Behavioral: Quit Center cessation program — Lifestyle modifications based on the Quit Center cessation program.

SUMMARY:
The goal of this clinical trial is to determine the success rate (efficacy) of a newly developed program to help smokers and vapers quit smoking. There will be no drugs of any nature involved, nor will there be any replacement addictions offered (ie; patches, gummies, etc.) It will also learn about the demographic profile of inbound participants. The main questions it aims to answer are:

Does the new program offer an improved success rate for smoking cessation? Does the program eliminate the need for long term "trigger" management? Does the program effectively diminish the anxiety that is normally associated with smoking cessation?

Participants will:

Attend a 1 hour group zoom session each week for the duration of the program (8 weeks).

Fill out an onboarding demographic questionnaire and exit demographic questionnaire.

Agree to a 6 month follow up questionnaire regarding their continued success/failure.

There are no physical meeting requirements. Participants can be located anywhere within the US.

DETAILED DESCRIPTION:
Participants will be sourced from within the United States. At this time, even though the program will be delivered online, the trial will be limited to US residents. It is anticpated that there will be a percentage of the participants that speak English as a second language, and therefore the Sponsor will also offer several sessions in Spanish. Participants MUST currently be smokers or vapers, as the basis of the test is to determine the anticipated success rate for participants to quit smoking.

The medical and emotional benefits of quitting smoking and ending nicotine addiction have been exhaustively tested in many previous studies and trials. The results of which are indisputable. This trial will not be assessing the ultimate benefits to ending the nicotine addiction. The primary purpose of this trial is to assess the efficacy of the holistic approach to quitting, and to gauge the program results against any currently extant methods. The program will instruct participants in ways to end their addiction to cigarettes and/or vaping, using their body's own natural abilities. It does NOT purport to be a medical solution, nor will any drugs be recommended or prescribed. There will also be NO reliance on other currently available medical/non-medical replacement therapies (ie; patches, gummies, hypnotism, prescription medication, etc,) and none of the personnel conducting any segment of the trial will be authorized to discuss or recommend any medical treatments whatsoever. The ultimate goal of the program is to completely eliminate the triggers that so often derail the effort to quit smoking.

Participants will step through an 8 week program, during which they will be shown ways to make incremental lifestyle changes that result in the cessation of the smoking addiction. The process is a holistic approach using the body's natural processes to eliminate anxiety. Additionally, each session will comprise groups of between 15-20 smokers. This will provide the "community" effect that will also add to the efficacy of the percentages.

ELIGIBILITY:
Inclusion Criteria:

1. must be addicted to nicotine either by cigarette or vaping
2. must have access to an internet connected device, laptop, or smartphone
3. must be 18 years old or older

Exclusion Criteria:

1. currently enrolled in any weight-loss program
2. currently enrolled in any behavioral modification program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study, although offered without geographical limitations, will be linited to United States residents
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Initial Cessation | 8 weeks
  percentage of participants that report quitting smoking by the end of the program

SECONDARY OUTCOMES:
Extended Cessation | 6 months
  percentage of participants that report staying quit for an extended time period
Permanent Cessation | 1 year
  percentage of participants that remain smoke free permanently

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rubino, Study Director — Quit Center LLC, Managing Member
Locations (1):
- QuitCenter.org, Beaufort, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be distributed. Aggregate data will be reported and will be available for other program's usage upon request to Quit Center LLC. Quit Center LLC reserves the right to limit the distribution of aggregate data.